CLINICAL TRIAL: NCT01823367
Title: Primary Prevention of Diabetes in Children and Mothers at Increased Risk: Encourage Healthy Families.
Brief Title: Encourage Healthy Families
Acronym: Encourage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: The JPB Foundation (Unknown); The YMCA of Greater Indianapolis (Unknown); Regenstrief Institute, Inc. (Other); Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, David Marrero, J.O Ritchey Professor of Medicine. Director, Diabetes Translational Research Center, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1207009188
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Gestational Diabetes Mellitus; Pre-diabetes
Keywords: type 2 diabetes mellitus prevention; gestational diabetes mellitus; pre-diabetes; lifestyle interventions; pediatric primary prevention of type 2 diabetes
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling mom only (Experimental): This intervention, delivered to groups of mothers only, builds upon the evidence-based curriculum used in the Diabetes Prevention Program (DPP) and incorporates into the curriculum detailed education regarding ways to help their children adopt healthier lifestyle behaviors.
  Interventions: Behavioral: Diabetes Prevention Program (DPP)
- Lifestyle counseling mom and child (Experimental): The second intervention is delivered to both mothers and children in separate groups using the same parent Diabetes Prevention Program (DPP) curriculum, but adds a group program for children that directly teach these children strategies for eating better and increasing physical activity.
  Interventions: Behavioral: Diabetes Prevention Program (DPP)

INTERVENTIONS:
Behavioral: Diabetes Prevention Program (DPP) — Diabetes Prevention Program (DPP): This is an evidence-based curriculum that has shown that it is possible to prevent or delay Type 2 Diabetes (T2D) in individuals if they keep a healthy weight, eat a nutritious diet, and stay physically active.

SUMMARY:
This study is a randomized intervention that will test two different approaches reflecting diverse levels of both intensity and cost, to achieving risk reduction of T2D. This will help address a critical question in the translation of primary prevention research into the public health: how much intensity (and thus cost) is required to achieve an effective outcome? In addition, the proposed study will address a critical need in diabetes prevention that has not received sufficient scholarly attention: the prevention of T2D in children. No studies of diabetes prevention similar in scope to the DPP have been performed in school-aged children; however, reducing childhood obesity is widely accepted as the primary pathway to decreasing the growing prevalence of T2D in the pediatric population.

DETAILED DESCRIPTION:
The proposed interventions will target mothers with a history of Gestational Diabetes (GDM), who gave birth to babies 9 pounds or greater, or who have prediabetes who are thus at very high risk for developing diabetes, and by virtue of their GDM/prediabetes, their children are also at high risk. Because of the genetic components involved, all children born by a woman afflicted with gestational diabetes mellitus or prediabetes have elevated risk of developing Type 2 Diabetes. This first intervention builds upon the evidence-based curriculum used in the DPP and incorporates into the curriculum detailed education regarding ways to help their children adopt healthier lifestyle behaviors. It will be delivered in groups of mothers only at community sites using trained laypeople. The second intervention will use the same parent curriculum, but adds a group program for children that teach them (directly) strategies for eating better and increasing physical activity. This program will be delivered to both mothers and children in separate groups. The group sessions will take place at the same time and in the same location by a trained facilitator.

ELIGIBILITY:
Inclusion Criteria:

* Adult females, age 18 or greater
* Body-mass index of ≥ 25 kg/m2
* Is a biological mother to a child between 8 and 15 years of age (child must live with biological mom)
* Is a biological mother with past diagnosis or history of gestational diabetes, prediabetes or gave birth to a child who weighed 9 pounds or greater at delivery
* Child, ages 8 to 15 years, to biological mother meeting inclusion criteria for Adult Females

Exclusion Criteria:

* Biological mother or biological child with diagnosis of Type 1 or 2 Diabetes Mellitus
* Biological mother or biological child with current A1c > 6.5%
* Biological mother or biological child current casual capillary blood glucose > 220mg/dl
* Biological mother or biological child with uncontrolled hypertension (Systolic Blood Pressure (SBP) >180 mmHg or Diastolic Blood Pressure (DBP) >105 mmHg)
* Biological mother or biological child with heart attack, stroke, or transient ischemic attack in the past 6 months
* Biological mother or biological child with chest pain, dizziness, or fainting with physical exertion
* Biological mother or biological child with Chronic Obstructive Pulmonary Disease (COPD) or asthma requiring home oxygen
* Biological mother or biological child with cancer treatment in the last 5 years
* Biological mother or biological child with any other known condition that could limit ability to become physically active or limit life span to <5 years
* Biological mother or biological child with history of anti-diabetic medication use (oral agents or insulin) except during past gestational diabetes
* Biological mother or biological child with self-report of any other condition associated with disordered glucose metabolism (including but not limited to):pregnancy; Cushing's syndrome; acromegaly; pheochromocytoma; chronic pancreatitis
* Biological mother or biological child with conditions or behaviors likely to affect the conduct of the study (including but not limited to): any reported developmental problems, unable or unwilling to provide informed consent/assent, unable or unwilling to communicate with study staff or engage in learning activities

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2012-12; Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Changes in weight | 3, 6, and 12 months after the beginning of the assigned intervention program
  Weight taken during data collection visits

SECONDARY OUTCOMES:
Changes in diet | 3, 6, and 12 months after the beginning of the assigned intervention program
  Assessed by the Food Frequency Questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Overall Officials: David G Marrero, PhD., Principal Investigator — Inidana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Palmer KNB, Garr Barry VE, Marrero DG, McKinney BM, Graves AN, Winters CK, Hannon TS. Intervention Delivery Matters: What Mothers at High Risk for Type 2 Diabetes Want in a Diabetes Prevention Program-Results from a Comparative Effectiveness Trial. Diabetes Ther. 2020 Oct;11(10):2411-2418. doi: 10.1007/s13300-020-00891-1. Epub 2020 Aug 8. PMID 32770443
- [Derived] Hannon TS, Carroll AE, Palmer KN, Saha C, Childers WK, Marrero DG. Rationale and design of a comparative effectiveness trial to prevent type 2 diabetes in mothers and children: the ENCOURAGE healthy families study. Contemp Clin Trials. 2015 Jan;40:105-11. doi: 10.1016/j.cct.2014.11.016. Epub 2014 Nov 29. PMID 25457793